CLINICAL TRIAL: NCT05718531
Title: Coronary Artery Ectasia, Thrombotic Background and Efficacy of Various Anti Thrombotic Regimens.
Brief Title: Coronary Artery Ectasia, Efficacy of Various Anti Thrombotic Regimens.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hamed Mohamed, Cardiology Specialist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Anti-Thrombotics CAE
Record Dates: First submitted 2022-12-03; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm | interventions — Rivaroxaban; Clopidogrel; Tablets; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- acute coronary syndrome group1 (Active Comparator): 50 patients will have triple therapy (Aspirin,75 mg once daily, clopidogrel 75 mg once daily, and Rivaroxaban 2.5mg BID) prescribed for 3 month, then clopidogrel and Rivaroxaban for the following 9 months.
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet twice daily; Drug: Clopidogrel 75 Mg Oral Tablet
- acute coronary syndrome group 2 (Active Comparator): 50 patients will be on Aspirin 75mg once daily, clopidogrel 75mg once daily for 1 year.
  Interventions: Drug: Clopidogrel 75 Mg Oral Tablet; Drug: Aspirin tablet 75 mg
- chronic coronary syndrome group 1 (Active Comparator): 33 patients with prescribed aspirin 75 mg once daily and Rivaroxaban 2.5 mg BID N.B: Patients with stents placement within a year will be excluded from this group
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet twice daily; Drug: Aspirin tablet 75 mg
- chronic coronary syndrome group 2 (Active Comparator): 33 patients with clopidogrel 75 mg once daily and Rivaroxaban 2.5mg BID
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet twice daily; Drug: Clopidogrel 75 Mg Oral Tablet
- chronic coronary syndrome group 3 (Active Comparator): 34 patients with aspirin 75 mg once daily and clopidogrel 75 mg once daily.
  Interventions: Drug: Clopidogrel 75 Mg Oral Tablet; Drug: Aspirin tablet 75 mg

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet twice daily — effect of rivaroxaban 2.5 mg twice daily on MACE and quality of life in coronary artery ectasia patients.
  Arms: acute coronary syndrome group1; chronic coronary syndrome group 1; chronic coronary syndrome group 2
Drug: Clopidogrel 75 Mg Oral Tablet — Used as control group in 2nd arm and 5th arm
  Arms: acute coronary syndrome group 2; acute coronary syndrome group1; chronic coronary syndrome group 2; chronic coronary syndrome group 3
Drug: Aspirin tablet 75 mg — Used as control group in 2nd arm and 5th arm
  Arms: acute coronary syndrome group 2; chronic coronary syndrome group 1; chronic coronary syndrome group 3

SUMMARY:
1. To evaluate short and intermediate clinical outcome of different anti-thrombotic regimens on major adverse cardiac events (MACE) and quality of life in coronary artery ectasia patients.
2. To evaluate role of P-selectin as a marker of cardiovascular risk in coronary artery ectasia.

DETAILED DESCRIPTION:
Coronary artery ectasia (CAE) is the diffuse dilatation of coronary artery. It is defined as a dilatation with a diameter of 1.5 times the adjacent normal coronary artery . Its prevalence ranges from 1.2%-4.9% with male to female ratio of 3:1.

CAE is more common in males. Hypertension is a risk Factor. Interestingly, patients with Diabetes Mellitus (DM) have low incidence of CAE. This may be due to down regulation of matrix metalloproteinase (MMP) with negative re-modelling in response to atherosclerosis. Smoking appears to be more common in patients with CAE than in those with coronary artery disease (CAD).

Treatment for CAE is a controversial topic, as there is lack of clinical trials and standardized guidelines, Current options include:

1. aggressive risk-factor modification
2. Management of the coronary artery disease if obstructive lesions are found. Anti-platelet therapy with aspirin has been suggested for all CAE patients since most have coexistent coronary artery obstructive lesions and high likelihood of developing a myocardial infarction (MI). There have not been any prospective random studies evaluating the role of adenosine diphosphate inhibitors as part of therapy.

Considering anticoagulation therapy to prevent coronary thrombus formation has been a debatable topic due to limited randomized trials.it was strongly suggested to use warfarin as the basic treatment for achieving long-term anticoagulation in one study.

Efficacy and safety of novel oral anti-coagulants (NOACs) are superior to warfarin in patients with non-valvular atrial fibrillation, By searching the literature, there are few cases of the application of NOACs in coronary ectasia.

Rivaroxaban has been showed to reduce ischemic events and cardiovascular mortality along with a higher risk for bleeding in Subjects with Acute Coronary Syndrome (ACS) suggested by the Anti-Xa therapy to lower cardiovascular events in addition to standard therapy in subjects with acute coronary syndrome-thrombolysis in myocardial infarction 51 trial on a background of clopidogrel treatment.

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with coronary artery ectasia either associated with obstructive or non-obstructive coronary artery disease after undergoing coronary angiography at cath. lab, cardiology department, Assiut university heart hospital, Assiut university.

Exclusion Criteria:

1. Atrial fibrillation
2. Left ventricular thrombus
3. severe Valvular heart disease.
4. Mechanical valve prothesis
5. Crusade score ≥ 41 (high - very high risk)
6. deep venous thrombosis, pulmonary embolism
7. renal failure stage IV-V.
8. known malignancy
9. Evidence of acute or chronic infection (by history or clinical examination).
10. History of systemic inflammatory or autoimmune disease.
11. History of any clinically significant endocrine, hematologic, respiratory, or metabolic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1 year
  Major adverse cardiac events occurence
P selectin marker | 1 year
  Correlation of P selectin marker with the severity of the disease.

SECONDARY OUTCOMES:
Bleeding risk | 1 year
  Bleeding events occurence

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy S. Mohammad, MD, Study Chair — Assiut University; Mahmoud A. Abdallah, MD, Study Director — Assiut University; Aly M. Tohamy, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Ramappa P, Kottam A, Kuivanemi H, Thatai D. Coronary artery ectasia--is it time for a reappraisal? Clin Cardiol. 2007 May;30(5):214-7. doi: 10.1002/clc.20002. PMID 17492685
- [Background] Doi T, Kataoka Y, Noguchi T, Shibata T, Nakashima T, Kawakami S, Nakao K, Fujino M, Nagai T, Kanaya T, Tahara Y, Asaumi Y, Tsuda E, Nakai M, Nishimura K, Anzai T, Kusano K, Shimokawa H, Goto Y, Yasuda S. Coronary Artery Ectasia Predicts Future Cardiac Events in Patients With Acute Myocardial Infarction. Arterioscler Thromb Vasc Biol. 2017 Dec;37(12):2350-2355. doi: 10.1161/ATVBAHA.117.309683. Epub 2017 Oct 19. PMID 29051141
- [Background] Khedr A, Neupane B, Proskuriakova E, Jada K, Kakieu Djossi S, Mostafa JA. Pharmacologic Management of Coronary Artery Ectasia. Cureus. 2021 Sep 8;13(9):e17832. doi: 10.7759/cureus.17832. eCollection 2021 Sep. PMID 34660041
- [Background] Pranata R, Yonas E, Chintya V, Alkatiri AA. Is Anticoagulant Necessary in Patients with Coronary Artery Ectasia Presenting with Acute Coronary Syndrome? A Systematic Review of Case Reports. Int J Angiol. 2019 Dec;28(4):231-236. doi: 10.1055/s-0039-1692706. Epub 2019 Jun 28. PMID 31787821
- [Background] Oldridge N, Hofer S, McGee H, Conroy R, Doyle F, Saner H; (for the HeartQoL Project Investigators). The HeartQoL: Part I. Development of a new core health-related quality of life questionnaire for patients with ischemic heart disease. Eur J Prev Cardiol. 2014 Jan;21(1):90-7. doi: 10.1177/2047487312450544. Epub 2012 Jul 20. PMID 22822179
- [Background] Oldridge N, Hofer S, McGee H, Conroy R, Doyle F, Saner H; (for the HeartQoL Project Investigators). The HeartQoL: part II. Validation of a new core health-related quality of life questionnaire for patients with ischemic heart disease. Eur J Prev Cardiol. 2014 Jan;21(1):98-106. doi: 10.1177/2047487312450545. Epub 2012 Jul 20. PMID 22822180